CLINICAL TRIAL: NCT01800006
Title: XANTUS-EL, Xarelto® on Prevention of Stroke and Noncentral Nervous System Systemic Embolism in Patients With Non-valvular Atrial Fibrillation in Eastern EU, Middle East, Africa (EMEA) and Latin America (LATAM): A Non-interventional Study
Brief Title: Xarelto for Prevention of Stroke in Patients With Atrial Fibrillation in Latinamerica and EMEA Region
Acronym: XANTUS-EL
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16691; XA1206 (Other: Company internal)
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Observation; Stroke; Embolism
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Embolism | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Patients with non-valvular atrial fibrillation who are prescribed Rivaroxaban under routine treatment conditions to prevent stroke or non-central nervous system systemic embolism. Decision regarding dose and duration of treatment made at the discretion of the attending investigator.

SUMMARY:
This international study is a prospective noninterventional observational cohort study of patients with non-valvular atrial fibrillation who are prescribed rivaroxaban under routine treatment conditions to prevent stroke or non-central nervous system systemic embolism. Patients will be followed up for 1 year or until 30 days after end of rivaroxaban therapy in case of therapy was discontinued earlier than 12 months. Serious adverse events will be followed up adequately. Laboratory values (e.g., Hb, HCT, haemoccult) should be documented for each point in time they were measured.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ 18 years of age with a diagnosis of non-valvular atrial fibrillation who start treatment with rivaroxaban to prevent stroke or non-CNS systemic embolism, and who consent to participate in the study.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation who are prescribed rivaroxaban under routine treatment conditions to prevent stroke or noncentral nervous system systemic embolism.
Sampling Method: Probability Sample
Enrollment: 2101 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2016-01-16 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Adjudicated major bleeding events | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Safety variables will be summarized using descriptivestatistics based on adverse events collection | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
All cause mortality | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later

SECONDARY OUTCOMES:
Adjudicated symptomatic thromboembolic events | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Non-major bleeding, collected as SAEs or non-serious AEs and defined as all bleeding events that do not fall in the category of major bleedings | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Treatment satisfaction | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Adverse events rates in the different AF risk factor categories | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Persistence with rivaroxaban treatment | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Reasons for switch of rivaroxaban treatment | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Reasons for interruption of rivaroxaban treatment | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Healthcare resource | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
  Number of healthcare professional visits and hospitalizations due to anticoagulation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (17):
- Many Locations, Argentina
- Many Locations, Azerbaijan
- Many Locations, Bahrain
- Many Locations, Chile
- Many Locations, Colombia
- Many Locations, Egypt
- Many Locations, Georgia
- ManyLocations, Jordan
- Many Locations, Kazakhstan
- Many Locations, Kenya
- ManyLocations, Lebanon
- Many Locations, Mexico
- Many Locations, Russia
- ManyLocations, Saudi Arabia
- Many Locations, United Arab Emirates
- Many Locations, Uruguay
- Many Locations, Venezuela

REFERENCES:
- [Derived] Kirchhof P, Haas S, Amarenco P, Turpie AGG, Bach M, Lambelet M, Hess S, Camm AJ. Causes of death in patients with atrial fibrillation anticoagulated with rivaroxaban: a pooled analysis of XANTUS. Europace. 2024 Jul 2;26(7):euae183. doi: 10.1093/europace/euae183. PMID 38941511
- [Derived] Kirchhof P, Radaideh G, Kim YH, Lanas F, Haas S, Amarenco P, Turpie AGG, Bach M, Lambelet M, Hess S, Camm AJ; Global XANTUS program Investigators. Global Prospective Safety Analysis of Rivaroxaban. J Am Coll Cardiol. 2018 Jul 10;72(2):141-153. doi: 10.1016/j.jacc.2018.04.058. PMID 29976287